CLINICAL TRIAL: NCT06869304
Title: Examining the Effect of Steep Trendelenburg Position on Neurocognitive Functions With MoCA Test in Robotic-assisted Radical Prostatectomy Surgeries.
Brief Title: The Effect of Steep Trendelenburg Position on Neurocognitive Functions in Robotic Radical Prostatectomy Cases
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Assoc. Prof, Ankara City Hospital Bilkent
Other Study IDs: TABED2-24-570
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Neurocognitive Disorder; Robotic Assisted Laparoscopic Radical Prostatectomy; Near Infrared Spectroscopy
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Montreal Cognitive Assessment — Preoperative and postoperative MoCA test scores

SUMMARY:
The aim of this study is to evaluate the effects of the steep Trendelenburg position in robotic prostatectomy cases, where anesthesia depth is monitored using BIS and cerebral perfusion is tracked with NIRS, and to determine the incidence of neurocognitive dysfunction using the MoCA test in the postoperative period.

Steep Trendelenburg position and CO₂ pneumoperitoneum during robotic radical prostatectomy lead to significant changes in intracranial pressure and cerebral oxygenation, which may contribute to postoperative neurocognitive dysfunction (POCD). Monitoring anesthesia depth with Bispectral Index (BIS) and cerebral perfusion with Near-Infrared Spectroscopy (NIRS) may help detect early neurocognitive changes, and MoCA test assessments will reveal a measurable decline in cognitive function postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* ASA II-III risk score
* Patients scheduled for robotic radical prostatectomy
* Patients who voluntarily agree to participate

Exclusion Criteria:

* Age < 65 years
* History of neurological or psychiatric disorders
* Inability to undergo robotic surgery
* Conversion to open prostatectomy during surgery
* Patients who do not consent to participate

Ages: 65 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 65 years and older with ASA II-III risk scores, undergoing robotic radical prostatectomy
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
MoCA | preoperatively
  Preoperative MoCA test scores
MoCA | day 1
  postoperative MoCA test scores

SECONDARY OUTCOMES:
NIRS | intraoperatively
  NIRS values (right & left)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided